CLINICAL TRIAL: NCT03564561
Title: Clinical and Molecular Aspects of Adult Onset Pompe Disease: a Natural History Study
Brief Title: Natural History of Pompe Disease
Acronym: POMPE
Status: Recruiting | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: P160405J; 2017-A02458-45 (Registry Identifier: N° ID RCB)
Record Dates: First submitted 2018-03-27; First posted 2018-06-21 (Actual); Last update posted 2024-04-08 (Actual); Status verified 2024-04

CONDITIONS: Glycogen Storage Disease Type II, Adult
Keywords: glycogen storage disease type II, adult; Pompe disease; clinical evolution; molecular evolution; follow-up; c.-32-13T>G mutation; antisense oligonucleotide treatment; in vitro
MeSH Terms: conditions — Glycogen Storage Disease Type II

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood, urine, skeletal muscle biopsy, skin biopsy:
  1. Blood for serum markers, DNA and white blood cell culture (lymphoblastoid cell line).
  2. Skeletal muscle biopsy for histology, RNA and protein analysis, myoblast culture.
  3. Skin biopsy for RNA and protein analysis, fibroblast culture.
  4. Urine for biomarker analysis.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The project is a prospective study in which patients affected by adult-onset Pompe disease with c.-32-13T>G mutation in the GAA gene will be followed-up during two years to describe the natural history using clinical, imaging, histological and molecular parameters.

Secondary objectives are:

* To identify biomarkers for assessing efficacy of future therapies based on correcting aberrant alternative splicing in Pompe patients with c.-32-13T>G mutations.
* To determine effectiveness of antisense oligonucleotide chemistries to restore full length GAA transcripts, GAA protein and GAA enzyme activity in fibroblasts and myoblasts obtained from skin and muscle biopsies as well as leucocytes of Pompe patients with c.-32-13T>G mutations.

DETAILED DESCRIPTION:
Study aim:

The principal objective of the study is to find biomarkers and clinical criteria that correlate with the disease progression.

Methods:

Clinical information will be obtained according to a pre-defined protocol including six visits: screening visit, visit at baseline, visits at 6 months, 12 months, 18 months and 24 months.

At visits following tests will be performed:

Respiratory assessment (including clinical assessment using the Borg scale, identification of clinical signs of alveolar hypoventilation, documentation of the daily duration on and off mechanical ventilation, spirometry, determination of lung volumes and slow vital capacity, peak cough flow, blood gazes, measurement of maximal inspiratory and expiratory pressures during the Müller maneuver, sniff nasal inspiratory pressure, mouth inspiratory pressure, twitch mouth pressure, esophageal and transdiaphragmatic pressures during voluntary respiration and following magnetic stimulation of diaphragmatic nerves, optoelectronic measurement of abdominal contribution to vital capacity, inspiratory capacity and tidal volume, measure of diaphragm mobility using ultrasound, sleep studies using polysomnography for non-ventilated patients and oximetry for patients using non-invasive mechanical ventilation, coupled with ECG recording).

Motor assessment (including the MFM motor function measure scale, timed 10 meters run/walk test, timed test for standing up from sitting positions, timed test for standing up from supine position, time taken to climb 4 stairs, 6-minute walk test, three-dimensional analysis of walk, quadriceps muscle strength assessed following magnetic stimulation of femoral nerve, EMG).

Assessment of body composition (including determination of lean mass, body mass index and bone mineral density by dual X-ray absorptiometry).

Assessment of skeletal muscle structure using whole body magnetic resonance imaging.

Assessment of heart function using heart echography and ECG. Assessment of live quality (including "Rotterdam handicap scale", "Rasch-built Pompe-specific Activity (R-Pact) scale " and EQ5D-5L questionnaires).

Biomaterial collection of biomarker analysis (including dosing serum CPK, GPT and GOT, GAA mutational analysis of both alleles, biobanking of serum, DNA and urine, muscle biopsy for histological analysis, quantification of exon 2 alternative splicing and residual GAA enzyme activity, myoblast culture for quantification of alternative splicing and residual GAA enzyme activity, muscle biopsy and myoblast culture biobanking, skin biopsy for quantification of alternative splicing and residual GAA enzyme activity, fibroblast cultures for quantification of alternative splicing and residual GAA enzyme activity, biobanking of fibroblasts).

In vitro treatment of myoblasts and fibroblasts with antisense oligonucleotide chemistries and quantification of restoration of normal splicing, GAA protein and GAA enzyme activity.

All data collect will be introduced in a database and afterwards statistically analyzed.

Expected results:

To determine exact natural history of Pompe disease, to identify biomarkers useful to follow-up the progression of Pompe disease and for quantifying therapy effects of future therapies that aim at restoring a normal splicing in patients with c.-32-13T>G mutations.

Funding:

This project is funded by the French Agence National de la Recherche, the French Direction Générale de l'Offre de Soins and the Acid Maltase Deficiency Association.

ELIGIBILITY:
Inclusion Criteria:

* Pompe disease Patient with c.-32-13T>G mutation in at least one allele of GAA gene.
* Ambulating patient : six-minute walk test distance > 50 m.
* Patient aged between 18 and 80 years.
* Informed consent signed par patient.
* Patient covered by a health insurance.

Exclusion Criteria:

* Invasive mechanical ventilation
* Pregnant woman
* Presence of comorbidity, in particular preexisting diseases like chronic infectious diseases (VIH infection, hepatitis or others), asthma, malignant tumour, hematologic diseases
* Patient who participate in another clinical trial
* Life expectancy < 12 months
* Unable to understand instructions and restraints of the study

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients between 18 and 80 years with adult-onset Pompe disease who carry the common c.-32-13T>G mutation of GAA gene, treated or not by Myozyme.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2019-06-07 (Actual); Primary Completion 2033-03 (Estimated); Study Completion 2033-03 (Estimated)

PRIMARY OUTCOMES:
The Six-Minute Walk Test | At baseline
The Six-Minute Walk Test | at 6 months
The Six-Minute Walk Test | at 12 months
The Six-Minute Walk Test | at 18 months
The Six-Minute Walk Test | at 24 months

SECONDARY OUTCOMES:
Moter assessment: quadriceps strength | At baseline, at 6, 12, 18 and 24 months
  Quadriceps muscle strength assessed following magnetic stimulated of femoral nerve.
Moter assessment: : the MFM moter function measure scale | At baseline, at 6, 12, 18 and 24 months
  Measurement of motor function by MFM (Motor Function Measure) scale.
Moter assessment: timed 10 meters run/walk test | At baseline, at 6, 12, 18 and 24 months
  Time for a 10-meter walk.
Moter assessment: timed test for standing up from sitting position | At baseline, at 6, 12, 18 and 24 months
  Time for getting up from a chair.
Moter assessment: timed test for standing up from supine position | At baseline, at 6, 12, 18 and 24 months
  Time for getting up from decubitus position.
Moter assessment: time taken to climb 4 stairs | At baseline, at 6, 12, 18 and 24 months
  Time for climbing 4 stairs.
Moter assessment: three-dimensional analysis of walk | At baseline, at 6, 12, 18 and 24 months
  3D analysis of walking.
Moter assessment: 6-minute walk test | At baseline, at 6, 12, 18 and 24 months
  The 6-minute walk test.
Body composition | At baseline, 12th and 24th months
  Osteodensitometry.
Body composition | At baseline, 12th and 24th months
  Body composition (ratio lean mass / fat mass) measure by dual-energy X-ray absorptiometry.
Body composition | At baseline, 12th and 24th months
  Body Mass Index (BMI).
Evaluation of skeletal muscle by MRI imaging | At baseline, 12th and 24th months
  Whole-body muscle MRI protocol :
  * Short tau inversion recovery (STIR).
  * T2-axial and coronal 3D.
  * IDEAL IQ.
Respiratory parameters: dyspnea using Borg scale | At baseline, at 6, 12, 18 and 24 months
  Evaluation of dyspnea using Borg scale.
Respiratory assessment: alveolar hypoventilation identification | At baseline, at 6, 12, 18 and 24 months
  Identification of clinical signs of alveolar hypoventilation.
Respiratory parameters: daily duration of non-ventilation for ventilated patients | At baseline, at 6, 12, 18 and 24 months
  Daily duration of non-ventilation for ventilated patients.
Heart function assessment | At baseline, at 6, 12, 18 and 24 months
  Assessment of heart assessment using heart echography
Heart function assessment | At baseline, at 6, 12, 18 and 24 months
  Assessment of heart assessment using ECG
Quality of life assessment | At baseline
  Evaluate by Questionnaire EQ5D-5L.
Quality of life assessment | At baseline
  Evaluate by Rotterdam handicap scale.
Quality of life assessment | At baseline
  Evaluate by Rasch-built Pompe-specific activity (R-Pact) scale.
Histological features | At baseline
  Histological study by using muscular biopsy culture with Periodic acid-Schiff stain and H&E stain.
Genotype | At baseline
  Determination of patient's GAA genotypes on blood sample.
Molecular and biochemical parameters: muscular biopsy | At baseline
  Muscular biopsy:
  Quantification of alternative splicing and residual enzymatic activity of acid alpha-glucosidase (GAA) of Pompe patient with c.-32 -13T>G mutation of GAA gene.
Molecular and biochemical parameters: cutaneous biopsy | At baseline
  Cutaneous biopsy:
  Quantification of alternative splicing and residual enzymatic activity of acid alpha-glucosidase (GAA) of Pompe patient with c.-32 -13T>G mutation of GAA gene.
Biomarkers | At baseline
  Blood sample (serum):
  Dosing of CPK, GPT and GOT level in serum.

CONTACTS AND LOCATIONS:
Overall Officials: Helge Amthor, MD, PhD, Principal Investigator — Hôpital Raymond Poincaré; Pascal Laforêt, MD, PhD, Study Director — Hôpital Raymond Poincaré
Locations (1):
- Hôpital Raymond Poincaré, Garches, Hauts-de-Seine, France

IPD SHARING:
Plan to Share IPD: No